CLINICAL TRIAL: NCT00610805
Title: Cardiology Prevention Trial in Systemic Lupus Erythematosus
Brief Title: Cardiology Prevention in Systemic Lupus Erythematosus (SLE)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Arthritis Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Jennifer Elliott, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO07050181
Record Dates: First submitted 2008-01-24; First posted 2008-02-08 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; lupus; cardiovascular; IMT; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants randomized to this arm (n=15) will be followed by Preventive Cardiology and will have appropriate goal oriented interventions on their risk factor levels for 2 years.
  Interventions: Other: Preventive Cardiology
- 2 (Other): Participants randomized to this arm (n=15) will receive usual care. The PI will send a letter of all testing results to their primary care physician. No standard care will be withheld.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Preventive Cardiology — Patients will receive those interventions recommended by the Preventive Cardiologist. This may include: exercise, electrocardiogram, specialized blood testing, blood pressure monitoring, nutrition counseling, smoking cessation counseling, and pharmacotherapy for hypercholesterolemia, hypertension, and blood sugar abnormalities.
  Arms: 1
Other: Usual Care — Participants will receive usual care per their primary care physician.
  Arms: 2

SUMMARY:
We propose a feasibility study of aggressive CV risk factor management directed by preventive cardiology compared to usual care. We will determine: 1) the efficacy of a preventive cardiology program compared to usual care in slowing the progression of carotid IMT and plaque, and 2) the effect of a preventive cardiology program versus usual care at achieving CV risk factor target goals.

We hypothesize Lupus patients randomized to the preventive cardiology program will have less cardiovascular progression over two years than those lupus patients who are given standard care for cardiovascular risk, defined by carotid intima-media thickness and plaque.

DETAILED DESCRIPTION:
We will recruit 30 eligible patients from the Lupus Center of Excellence outpatient clinic. Patients will either be randomized into a preventive cardiology program for aggressive treatment, or randomized to usual care (1:1 ratio) in a single-blinded, randomized trial of 24 months duration. In this feasibility trial we hope to identify and refine any limitations in anticipation of designing a larger, randomized intervention study.

For both arms of the study, at baseline, 6 month, 12 month, 18 month, and 24 month visits (5 visits in total) all patients will be seen by Dr. Elliott, Principal Investigator. Visits will include an interview, fasting laboratory tests completion of questionnaires regarding demographics, socioeconomic status, health status, and risk factors (traditional, inflammatory, and lupus-specific). Dr. Elliott will perform the physical examinations on all patients and complete the lupus-specific disease activity and damage questionnaires. At the Baseline visit, 12-month visit, and 24 24-month visits, all patients will have a carotid ultrasound.

Cohort 1: Preventive Cardiology Program arm: Above and beyond the standard care, which is listed below, the patients in this arm will be aggressively treated by the cardiologist. As deemed prudent, the following may be prescribed: antihypertensives, lipid reducing agents, anti-platelets, further cardiac testing, and behavioral modifications. No standard care treatment will be withheld.

Cohort 2: Standard Care arm: The PI will send a letter of all testing results to their designated PCP. No standard care treatment will be withheld.

ELIGIBILITY:
Inclusion Criteria:

1. Definitive diagnosis of SLE
2. >18 years of age
3. Followed by rheumatologists (not the investigator, Dr. Elliott) at the Lupus Center of Excellence
4. Informed consent signed
5. Effective form of birth control

Exclusion Criteria:

1. Prior cardiovascular disease history (MI, coronary angioplasty, coronary artery bypass graft, abnormal coronary angiography, abnormal nuclear or treadmill stress test)
2. Prior evaluation by preventive cardiology
3. Active cardiac issues
4. Pregnancy, breastfeeding, or anticipating pregnancy in the next 2 years

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The efficacy of a preventive cardiology program compared to usual care in slowing the progression of carotid IMT and plaque | 2 years
The effect of a preventive cardiology program versus usual care at achieving CV risk factor target goals. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Elliott, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Lupus Center of Excellence, Magee Womens Hospital, 300 Halket St, Suite 1750, Pittsburgh, Pennsylvania
  - Clinical and Translational Research Center (CTRC), Montefiore Hospital, 6NE, 200 Lothrop St., Pittsburgh, Pennsylvania